CLINICAL TRIAL: NCT02047539
Title: Randomized Controlled Trial of Aspirin vs Placebo in the Treatment of Patients With the Clinical Risk Syndrome for Psychosis
Brief Title: Randomized Controlled Trial of Aspirin vs Placebo in the Treatment of Pre-psychosis
Status: Terminated | Phase: Early Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Health Services Research
Other Study IDs: 1401013288
Record Dates: First submitted 2014-01-24; First posted 2014-01-28 (Estimated); Last update posted 2021-05-17 (Actual); Status verified 2021-05

CONDITIONS: Clinical High Risk for Psychosis
MeSH Terms: interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1000 mg/day aspirin (Experimental): 1000 mg/day aspirin
  Interventions: Drug: Aspirin
- sugar pill (Placebo Comparator): sugar pill
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Aspirin — 1000 mg/day of aspirin 1000 mg/day of sugar pill
  Arms: 1000 mg/day aspirin
Drug: Placebo
  Arms: sugar pill

SUMMARY:
The primary objective of this study is to determine whether aspirin is effective in alleviating symptoms of the clinical high risk (CHR) syndrome for psychosis. The investigators further aim to determine whether it may delay or prevent the onset of psychosis in those currently experiencing CHR symptoms. As secondary measures the investigators aim to collect laboratory studies of inflammation markers and genetic samples to determine whether certain genetic profiles correlate with risk for psychosis, or response to aspirin treatment.

DETAILED DESCRIPTION:
Patients will be randomly assigned to either active treatment (aspirin) or placebo.

ELIGIBILITY:
Inclusion Criteria:

* Age 19 - 35
* Must have a SIPS interview
* CHR subjects must meet at least one of 3 CHR syndromes defined by SIPS
* Must demonstrate adequate decisional capacity

Exclusion Criteria:

* Under age of 19
* Have pre-existing gastrointestinal disease, heart disease
* Have kidney disease
* Taking non-steroidal anti-inflammatory medications
* Hypersensitive to NSAID (non-steroidal anti-inflammatory medications)
* Have coexisting unstable major medical illness
* Are pregnant or breastfeeding
* Consume more than 2 drinks of alcohol per day
* Have a blood clotting disorder
* Are taking ACE inhibitors, acetazolamide, anticoagulants, anticonvulsants, beta blockers, diuretics, methotrexate, oral hypoglycemic or uricosuric agents
* Have a history of substance abuse in past three moths or dependence in past 6 months

Ages: 19 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 1 (Actual)
Dates: Start 2015-01; Primary Completion 2021-03 (Actual); Study Completion 2021-03 (Actual)

PRIMARY OUTCOMES:
Scale of Prodromal Symptoms (SOPS) | 2 weeks
  Patients randomized to aspirin will improve significantly more on the SOPS total score than patients randomized to placebo
Scale of Prodromal Symptoms (SOPS) | 4 weeks
  Patients randomized to aspirin will improve significantly more on the SOPS total score than patients randomized to placebo
Scale of Prodromal Symptoms (SOPS) | 8 weeks
  Patients randomized to aspirin will improve significantly more on the SOPS total score than patients randomized to placebo
Scale of Prodromal Symptoms (SOPS) | 12 weeks
  Patients randomized to aspirin will improve significantly more on the SOPS total score than patients randomized to placebo

CONTACTS AND LOCATIONS:
Overall Officials: Scott W Woods, MD, Principal Investigator — Yale University
Locations (1):
- PRIME Research Clinic, New Haven, Connecticut, United States